CLINICAL TRIAL: NCT00244387
Title: A Multi-centre, Multi-national, Phase 3, Randomized, Double-blind, Double-dummy, 3- Arm Parallel Group, Placebo- and Pramipexole- Controlled Trial of the Efficacy and Safety of Rotigotine Patch in Subjects With Advanced Stage, Idiopathic Parkinson's Disease Who Are Not Well Controlled on Levodopa
Brief Title: Rotigotine Patch in Subjects With Advanced Stage, Idiopathic Parkinson's Disease Who Are Not Well Controlled on Levodopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0515
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2010-02

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: advanced stage idiopathic Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: SPM 962

SUMMARY:
Male and female patients aged ≥ 30 years with advanced stage idiopathic Parkinson's disease, not well controlled on existing levodopa will take part in a research study at approximately 82 sites in Europe, Israel, South Africa, Australia and new Zealand.

The purpose of the study is to evaluate the effectiveness, safety and tolerability of the rotigotine patch (SPM 962) at an individual patient's optimal dose for a period of 4 months

Each patient who qualifies and chooses to participate in the study will receive either rotigotine, pramipexole, or placebo at gradually increasing doses over a period of up to 7 weeks, and then maintain their optimal dose for 4 months.

The study clinic visits will include a medical history and physical exam, ECG, blood and urine sample collection, completion of various questionnaires, and completion of a diary to record the severity of their Parkinson's symptoms.

Patients who complete the study may enroll in an extension trial and receive active study drug.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage idiopathic Parkinson's disease

Exclusion Criteria:

* Well controlled on levodopa

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2004-03; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany

REFERENCES:
- [Result] Poewe WH, Rascol O, Quinn N, Tolosa E, Oertel WH, Martignoni E, Rupp M, Boroojerdi B; SP 515 Investigators. Efficacy of pramipexole and transdermal rotigotine in advanced Parkinson's disease: a double-blind, double-dummy, randomised controlled trial. Lancet Neurol. 2007 Jun;6(6):513-20. doi: 10.1016/S1474-4422(07)70108-4. PMID 17509486
- [Result] Pahwa R. Rotigotine skin patch for the treatment of fluctuating Parkinson's disease--how does it compare with pramipexole? Nat Clin Pract Neurol. 2007 Dec;3(12):656-7. doi: 10.1038/ncpneuro0632. Epub 2007 Sep 25. No abstract available. PMID 17895872
- [Result] Oertel W, LeWitt P, Giladi N, Ghys L, Grieger F, Boroojerdi B. Treatment of patients with early and advanced Parkinson's disease with rotigotine transdermal system: age-relationship to safety and tolerability. Parkinsonism Relat Disord. 2013 Jan;19(1):37-42. doi: 10.1016/j.parkreldis.2012.06.009. Epub 2012 Sep 3. PMID 22954721
- [Derived] LeWitt PA, Poewe W, Elmer LW, Asgharnejad M, Boroojerdi B, Grieger F, Bauer L. The Efficacy Profile of Rotigotine During the Waking Hours in Patients With Advanced Parkinson's Disease: A Post Hoc Analysis. Clin Neuropharmacol. 2016 Mar-Apr;39(2):88-93. doi: 10.1097/WNF.0000000000000133. PMID 26882318